CLINICAL TRIAL: NCT03852654
Title: A Novel 18F-DCFPyL PET-CT Scan for Diagnosis and Management of Prostate Cancer
Brief Title: 18F-DCFPyL PET-CT Scan and Prostate Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lida Jafari (U.S. Federal Agency)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor-Investigator, Lida Jafari, Nuclear Medicine Physician, VA Greater Los Angeles Healthcare System
Organization: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Jafari0001
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer Adenocarcinoma
Keywords: Prostate Cancer, PET CT scan, 18F-DCFPyL
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental)
  Interventions: Drug: 18F-DCFPyL

INTERVENTIONS:
Drug: 18F-DCFPyL — Subjects with biopsy proven prostate cancer, no prior local therapy, and:
  PSA ≥ 10 ng/dl, or Gleason Sum ≥ 4+3, or clinical stage ≥cT2c Staging by 99mTc-MDP or NaF PET bone scan, and Diagnostic CT (pelvis) or MRI will undergo 18F DCFPyL PET CT scan.

SUMMARY:
Primary Objective:

The primary objective of this study is to assess the efficacy of 18F-DCFPyL PET-CT for initial staging of prostate cancer in Veterans compared to conventional imaging (99mTc-MDP bone scan and Diagnostic CT or MRI). The primary clinical endpoint of our study is the percent of Veterans with prostate cancer in which the 18F-DCFPyL PET-CT identifies M1 disease at initial staging.

Secondary Objectives:

Frequency of the change in primary treatment plan after initial staging.

DETAILED DESCRIPTION:
This is a single arm Phase II clinical trial in Veterans with prostate cancer, no prior local therapy, who are at risk of having metastatic disease (PSA greater than 10, or Gleason Score greater than or equal to 4+3, or clinical stage greater than or equal to T2c). Veterans who are planned to undergo or have recently undergone conventional, routine care initial staging scans for prostate cancer (99mTc-MDP or NaF PET bone scan and diagnostic CT or MRI of pelvis) will also receive a 18F-DCFPyL PET-CT scan. The primary endpoint is the percent of Veterans with prostate cancer in which the 18F-DCFPyL PET-CT scan identifies evidence of M1 disease at initial staging.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and male.
2. Ability to understand the study and the willingness to sign a written informed consent document.
3. Histologically confirmed adenocarcinoma of the prostate.
4. PSA greater than 10, or Gleason ≥4+3, or clinical stage greater than or equal toT2c.
5. Plan to undergo (or have already undergone) routine care initial systemic staging with conventional imaging for prostate cancer.
6. Eastern Cooperative Oncology Group (ECOG) Performance score of 0 to 2.
7. No prior local therapy for prostate cancer (i.e., prostatectomy, radiotherapy, etc.).
8. Willing to comply with the procedural requirements of this protocol.

Exclusion Criteria:

1. Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection.
2. The subject has a condition or situation that, in the investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with subject's participation in the study.
3. Primary small cell carcinoma of the prostate.
4. Participation in this study significantly delay the scheduled standard of care therapy.
5. Weighs greater than 350 lbs., or unable to fit within the imaging gantry.
6. The subject undergone prior local therapy for prostate cancer (i.e. prostatectomy, radiotherapy, etc.).
7. Currently receiving androgen deprivation therapy (ADT) or anti-androgen? Previous use of ADT is allowed IF the subject has been off ADT or anti-androgen for 3 months or more.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2018-07-22 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
the percent of Veterans with prostate cancer in which the 18F-DCFPyL PET-CT identifies M1 disease at initial staging | 120 days

CONTACTS AND LOCATIONS:
Locations (1):
- VA Greater Los Angeles, Los Angeles, California, United States